CLINICAL TRIAL: NCT05157100
Title: Prospective, Open-label Clinical Study of Ingrezza (Valbenazine) for the Treatment of Cervical Dystonia
Brief Title: Clinical Study of Ingrezza (Valbenazine) for the Treatment of Cervical Dystonia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Orthopedic Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1002
Record Dates: First submitted 2021-11-30; First posted 2021-12-14 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Cervical Dystonia
MeSH Terms: conditions — Torticollis | interventions — valbenazine

STUDY DESIGN:
Intervention Model Description: Experimental
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Ingrezza (Experimental): Participants will receive Ingrezza orally once daily for 12 weeks.
  Interventions: Drug: Ingrezza Pill

INTERVENTIONS:
Drug: Ingrezza Pill — Participants will receive Ingrezza 40 mg and 80 mg tablets for 12 weeks.

SUMMARY:
Study of Ingrezza (Valbenazine) for the treatment of cervical dystonia.

DETAILED DESCRIPTION:
The study will be an open-label, prospective study. Patients with a diagnosis of cervical dystonia will undergo 4 weeks of baseline evaluation, followed by a 12-week treatment period. Subjects will be evaluated in-clinic every 4 weeks. Standardized assessments will be performed at these visits. Data will also be collected from wearable IMUs (inertial measurement units) and analyzed for improvements in involuntary, repetitive movements and postures.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients between 18 and 85 years of age (inclusive)
* A clinical diagnosis of cervical dystonia (ie, spasmodic torticollis) by investigator for at least six months
* Moderate to severe head tremor and/or dystonic posturing as judged by the investigator
* Stable Botulinum Toxin (Botox, Dysport, Xeomin, or Myobloc) therapy dosage for at least 3 months prior to baseline visit

Exclusion Criteria

* Tardive dyskinesia
* Predominant anterocollis
* Concomitant use of strong CYP3A4 inhibitors (i.e. itraconazole, ketoconazole, clarithromycin), digoxin, strong CYP2D6 inhibitors (i.e. paroxetine, fluoxetine, quinidine), monoamine oxidase inhibitors (i.e. isocarboxazid, phenelzine, selegiline)
* Myotomy or denervation surgery in the affected muscles (eg, peripheral denervation and/or spinal cord stimulation)
* Diagnosis of Myasthenia gravis, Lambert-Eaton syndrome, amyotrophic lateral sclerosis, or any other significant neuromuscular disease which might interfere with the trial
* Moderate to severe hepatic impartment as determined by a Child-Hugh Score ≥7
* Marked limitation on passive range of motion that suggests contractures or other structural abnormality, eg, cervical contractures or cervical spine syndrome
* Any conditions that may increase the risk associated with study participation or may interfere with the interpretation of study results and, in the judgment of the Investigator, would make the patient inappropriate for entry into this study
* Participation in another interventional study during participation in this study
* Pregnant or lactating females, or females of child-bearing potential not willing to use an acceptable method of contraception
* History of hypersensitivity to valbenazine or any components of INGREZZA.
* Is suicidal at screening as defined by below:

  1. According to the C-SSRS, he or she must not be actively suicidal at Visit 1 (Screening) or Visit 2 (Baseline) (including, an answer of "yes" to C-SSRS questions 4 or 5 [current or over the last 6 months]) and must not have attempted suicide in the 1 year prior to Visit 1 (Screening); OR
  2. The subject is actively suicidal in the Investigator's judgment

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-10-19 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Change in incidence of pain/spasm | 16 weeks
  Change in incidence rate of pain/spasm as measured by frequency and intensity in subjects prior to and during use of valbenazine as measured by Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS) and Inertial measurement unit (IMU). TWSTRS is a composite scale used to measure three aspects of CD: severity, disability, and pain. TWSTRS total score falls within the range of 0 to 85, where a higher score indicates a more severe condition.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Taylor, DO, PHD, Principal Investigator — principle investigator
Locations (1):
- The Orthopedic foundation, New Albany, Ohio, United States

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2021-09-06): https://cdn.clinicaltrials.gov/large-docs/00/NCT05157100/Prot_ICF_000.pdf